CLINICAL TRIAL: NCT05650684
Title: Factors Associated With Continuation of Exclusive Breastfeeding Until the Post-natal Visit
Acronym: PoursuitAllait
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_013_Poursuit-Allait
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Breastfeeding
Keywords: exclusive breastfeeding; postnatal visit; factors associated
MeSH Terms: conditions — Breast Feeding | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "exclusive breastfeeding" group: Women initiating exclusive breastfeeding after birth
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — continuation of exclusive breastfeeding until the post-natal visit (6 to 8 weeks after birth)

SUMMARY:
Breastfeeding promotes the health of mother and her child, and remains the reference in terms of infant nutrition. World Health Organization recommends exclusive breastfeeding for the first six months. This recommended duration is not respected in France with a median duration of breastfeeding in France at 3 months.

DETAILED DESCRIPTION:
The aim is to study factors associated with continuation of exclusive breastfeeding until the post-natal visit.

ELIGIBILITY:
Inclusion Criteria:

* primiparous and multiparous women
* women who have initiate breastfeeding
* women aged 18 and more
* agreeing to participate in the study

Exclusion Criteria:

* women whose newborn has been in intensive care unit
* women with a multiple pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Mother initiating exclusive breastfeeding after birth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
breastfeeding | Day 0
  number of women practicing or not exclusive breastfeeding until postnatal consultation (6 to 8 weeks after birth)